CLINICAL TRIAL: NCT02341573
Title: Effect of Experienced Chinese Herbal Formulas Based on Different Stages and Different Symptoms on Pediatric Asthma: a Single-blinded Randomized Controlled Trial
Brief Title: Experienced Chinese Herbal Formulas on Pediatric Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Yonghong Wang, Professor, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. 12401905500
Record Dates: First submitted 2014-12-31; First posted 2015-01-19 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Childhood Asthma
Keywords: Traditional Chinese Medicine; Randomized Controlled Trial
MeSH Terms: interventions — Leukotriene Antagonists; montelukast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chinese medicine group (Experimental): Children of chinese medicine group will be treated with experienced chinese herbal formula based on different stages and different symptoms.Patients at the acute stage of asthma will be given Shegan mixture ,at the remission stage, will be treated with Huangqi Bushen mixture-based formulation with modification according to their symptoms,10-30 mL , 2 times a day, for 3 months.
  Interventions: Drug: experienced chinese herbal formulas
- western medicine group (Active Comparator): Children of western medicine group will be treated with leukotriene receptor antagonist and a bronchial relaxant.Children at the acute stage of asthma will be treated with etinoline,twice a day for 7 days.At the remission stage, they will be given leukotriene receptor antagonist Singulair, once daily for 3 months.
  Interventions: Drug: leukotriene receptor antagonist and bronchial relaxant

INTERVENTIONS:
Drug: experienced chinese herbal formulas — At the acute stage of asthma :Shegan mixture ; At the remission stage:Huangqi Bushen mixture; 10-30 mL , 2 times a day, for 3 months.
  Other Names: Shegan mixture ,Huangqi Bushen mixture
  Arms: chinese medicine group
Drug: leukotriene receptor antagonist and bronchial relaxant — At the acute stage of asthma : etinoline,twice a day for 7 days; At the remission stage: Singulair, once daily for 3 months.
  Other Names: Singulair,etinoline,
  Arms: western medicine group

SUMMARY:
The purpose of this study is conducting a randomized, single blind, controlled intervention trial to observe the therapeutic effect of experienced chinese herbal formulas based on different stages and different symptoms in pediatric asthma.

DETAILED DESCRIPTION:
Pediatric bronchial asthma is a common disease that severely threatens physical and mental health of children. It's urgent to explore effective ways to alleviate the pain caused by asthma.

In our research, 160 asthmatic children are randomly divided into a Chinese medication group (80 cases) and a Western medication control group(80 cases). Patients in the Chinese medication group are treated with a series of experienced chinese herbal formulas, whereas the western medication control group received a leukotriene receptor antagonist and a bronchial relaxant. The Chinese medicine syndromes and western medicine symptoms are scored. Pulmonary function and asthma control test score will be applied in this study. We evaluate the situation of asthma from different aspects, including index of pulmonary function and score of asthma control test. Real-time PCR was used to determine the mRNA expression levels of some inflammatory mediators in peripheral.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they (a) were satisfying the above-mentioned diagnostic criteria with pediatric asthma and cough variation asthma, (b) aged 3-12 years, and (c) were with pattern of phlegm-heat obstruction and cold fluid-retention in lungs at the acute stage, or with pattern of lung-spleen deficiency and kidneyQideficiency at the remission stage of asthma based on traditional chinese medicine syndrome differentiation diagnosis.

Exclusion Criteria:

* Patients were excluded if they had congenital respiratory system diseases, tumors, immunodeficiency diseases, or cardiovascular diseases.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control Test Score | Baseline and 3 months
  We will measure the change in asthma control test scores between chinese medicine group and western medicine group.

SECONDARY OUTCOMES:
Change in mRNA expression levels of inflammatory mediators | Baseline and 3 months
  We will measure the change in mRNA expression levels of some inflammatory mediators in peripheral with Real-time PCR.
Change in some index of pulmonary function (PEF,FEV1,VT,etc.) . | Baseline and 3 months
  We will measure the change of some index of pulmonary function (PEF,FEV1,VT,etc.) .
Change in chinese medicine symptoms scores | Baseline and 3 months
  We will measure the Change in scores of chinese medicine symptoms(cough,expectoration,asthma attacks) according to the Traditional Chinese Medicine Guideline Scale: 0 - 3. 0 = None. 1 = Mild. 2 = Moderate. 3= Severe.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Y hong, professor, Study Chair — Children Hospital of Fudan University
Locations (1):
- Department of Chinese Traditional Medicine; Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China